CLINICAL TRIAL: NCT02984514
Title: Studies of Activity of Brown Adipose Tissue With Positron Emission Tomography Using the Tracer 18F-deoxy Glucose in Patients With Type 1 Diabetes
Brief Title: Brown Adipose Tissue in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per-Ola Carlsson (Other)
Responsible Party: Sponsor-Investigator, Per-Ola Carlsson, Professor, Senior consultant, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Dnr 2015/191
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Type 1 diabetes (Experimental): Positron emission tomography with tracer 18F-deoxy glucose
  Interventions: Radiation: Positron emission tomography with tracer 18F-deoxy glucose

INTERVENTIONS:
Radiation: Positron emission tomography with tracer 18F-deoxy glucose — Assessment of activity of brown adipose tissue with positron emission tomography using the tracer 18F-deoxy glucose

SUMMARY:
Brown adipose tissue has the capacity to consume large amounts of energy and has insulin-independent glucose uptake. The investigators have recently observed an inverse correlation between irisin levels and insulin needs of type 1 diabetes patients. Transplantation of brown adipose tissue to insulin-deficient rats normalized their blood glucose levels.

In this study 12 patients with long-standing type 1 diabetes (>10 years) and with variable exogenous insulin needs will be investigated for amount of brown adipose tissue with positron emission tomography using the tracer 18F-deoxy glucose.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years of age or more)
2. Type 1 diabetes diagnose for more than 10 years

Exclusion Criteria:

1. Ongoing pregnancy
2. Ongoing breast-feeding
3. BMI<19
4. BMI >30
5. P-creatinine <110 µmol/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-10; Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Activity of brown adipose tissue in correlation to exogenous insulin needs using the tracer 18F-deoxy glucose in positron emission tomography measurements | Assessment performed after more than 10 years of diagnosed type 1 diabetes

SECONDARY OUTCOMES:
Glucose uptake in muscle in correlation to exogenous insulin needs; assessment using the tracer 18F deoxy glucose in positron emission tomography measurements. | Assessment performed after more than 10 years of diagnosed type 1 diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden